CLINICAL TRIAL: NCT06962982
Title: Effect of Short Term Immersive VR Intervention With Exercises and Ergonomic Training on Neck Pain, Cervical ROM, Neck Endurance, Neck Disability and Work Productivity Among Computer Users.
Brief Title: This Study Explores How Short-term Immersive VR With Exercises and Ergonomic Training Can Reduce Neck Pain, Improve Movement, Strength, and Work Productivity in Computer Users Who Are at High Risk Due to Prolonged Screen Time and Poor Posture.
Acronym: VR ROM
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Gulf Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB-COHS-STD-9-Jan-2025
Record Dates: First submitted 2025-04-30; First posted 2025-05-08 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-04

CONDITIONS: Neck Pain; Neck Disability; Neck Endurance; Work Productivity; Cervical Range of Motion
Keywords: ergonomic training; neck pain; cervical ROM; neck endurance; neck disability; work productivity; computer users
MeSH Terms: conditions — Neck Pain | interventions — Exercise Therapy

STUDY DESIGN:
Intervention Model Description: participants will be randomly divided into two groups
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A - Therapeutic exercises and Ergonomic training. (Experimental): An initial ergonomic assessment of all the participants' workstation will be done using the Computer Workstation Self-Assessment Checklist to identify potential risk factors for neck pain and dysfunction. Numeric pain rating values, Neck muscle endurance, cervical range of motion, neck disability index and work productivity score will be measured and recorded for each participant.
  This group will receive therapeutic exercises including stretching and active exercises. Recommendations for adjustments to the chair, desk, and equipment layout would also be given to optimize comfort and efficiency and reduce neck pain due to improper workstation design. The session will last for 15 minutes. Follow up 2 days in a week over the 3-week period will be done to make necessary adjustments, and reinforce the ergonomic principles. All outcome measure will be attained again at the end of the 3 week period.
  Interventions: Behavioral: Therapeutic Exercises; Behavioral: Ergonomic Training
- Group B: Therapeutic exercises Ergonomic Training, and Immersive VR therapy. (Experimental): An initial ergonomic assessment of all the participants' workstation will be done using the Computer Workstation Self-Assessment Checklist to identify potential risk factors for neck pain and dysfunction. Numeric pain rating values, Neck muscle endurance, cervical range of motion, neck disability index and work productivity score will be measured and recorded for each participant.
  The participants of this group will be given all the trainings as Group A along with the addition of immersive VR. This task will be delivered through the Human XR device Oculus Quest 3. The VR module will involve participants to engage in targeted cervical movements (flexion, extension, rotation) to attain therapeutic objectives through visual cues. Group B will be given VR therapy for an additional 20 minutes. Follow up 2 days in a week over the 3-week period will be done for the participant to use the immersive VR mode. All outcome measure will be attained again at the end of the 3 week period.
  Interventions: Behavioral: Therapeutic Exercises; Behavioral: Ergonomic Training; Device: Human XR device - Oculus Quest 3

INTERVENTIONS:
Behavioral: Therapeutic Exercises — Therapeutic exercises including stretching and active exercises for neck and shoulder.
Behavioral: Ergonomic Training — Recommendations for adjustments to the chair, desk, and equipment to optimize comfort and efficiency and reduce unnecessary stress and loading on neck muscles.
Device: Human XR device - Oculus Quest 3 — Meta Quest 3 is a standalone virtual reality headset by Meta Platforms featuring a slimmer design, higher-resolution dual LCD displays, improved performance with the Snapdragon XR2 Gen 2 chip, and advanced mixed reality capabilities through color passthrough cameras and a depth sensor.
  Arms: Group B: Therapeutic exercises Ergonomic Training, and Immersive VR therapy.

SUMMARY:
The goal of this clinical trial is to learn if a short-term immersive Virtual Reality (VR) intervention, combined with exercises and ergonomic training, can help treat neck pain in computer users. It will also explore how safe and effective this approach is. The main questions it aims to answer are:

Does immersive VR with exercise and ergonomic training reduce neck pain and disability?

Does it improve cervical range of motion, neck muscle endurance, and work productivity?

Researchers will compare the effects before and after the intervention to see how well it works for managing neck pain in computer users.

Participants will:

Use immersive VR exercises and receive ergonomic training over a short period

Attend assessment sessions to measure pain, movement, endurance, and work productivity

Follow specific guidelines for posture and workplace adjustments during the study

ELIGIBILITY:
Inclusion Criteria:

1. Computer users of age 18 to 50 years old with history of more than 6 hours of screen time. (9)
2. Complaints of neck pain.

Exclusion Criteria:

1. Individuals having complains of vertigo
2. Radiating pain
3. Balance issues
4. Motion sickness
5. Recent cervical fractures/dislocations or whiplash injuries
6. Complaints of photosensitivity
7. Complaints of frequent headaches

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2025-05-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
The Numeric Pain Rating Scale | 3 weeks
  The Numeric Pain Rating Scale asks individuals to rate their pain intensity on a scale from 0 (no pain) to 10 (worst pain imaginable), with higher numbers indicating greater pain severity. The Numeric Pain Rating Scale (NPRS) demonstrates robust psychometric properties across multiple studies, making it a valuable tool for pain assessment in clinical practice. It exhibits excellent test-retest reliability, with coefficients ranging from 0.72 to 0.95 and intraclass correlation coefficients of 0.82 to 0.95 across various patient populations. Additionally, the NPRS is highly acceptable to patients due to its simplicity, can be administered verbally or in writing.
Cervical Range of Motion | 3 weeks
  Cervical range of motion (CROM) is a clinically critical outcome measure for assessing neck dysfunction, treatment efficacy, and rehabilitation progress. CROM measurments provide objective, quantifiable data to assess neck dysfunction severity, monitor rehabilitation progress, and evaluate treatment effectiveness, enabling clinicians to tailor interventions and predict recovery outcomes in patients with musculoskeletal or neurological conditions.

SECONDARY OUTCOMES:
The Neck Disability Index | 3 weeks
  The Neck Disability Index (NDI) is a validated, patient-reported outcome measure assessing neck pain-related disability across 10 domains, including daily activities, work, and sleep. It is scored from 0 (no disability) to 50 (complete disability). Widely used in clinical and research settings, it effectively tracks rehabilitation progress and treatment efficacy in conditions like neck pain and neck dysfunction.
Computer Workstation Ergonomics Self-Assessment Checklist | 3 weeks
  The Computer Workstation Ergonomics Self-Assessment Checklist is a reliable and practical tool that helps individuals evaluate their workstation setup, including seating, monitor placement, and input device positioning. It promotes user awareness of ergonomic principles and encourages healthy work habits, such as taking regular breaks. Widely used in both clinical and workplace settings, this checklist supports the prevention of musculoskeletal discomfort by guiding users toward effective ergonomic adjustments.
Work Productivity and Activity Impairment Questionnaire | 3 weeks
  The Work Productivity and Activity Impairment (WPAI) Questionnaire is a validated 6-item tool measuring health-related productivity loss, assessing absenteeism (work time missed), presenteeism (reduced effectiveness), overall work impairment, and activity limitations over seven days. It effectively distinguishes productivity outcomes by disease severity and its standardized scoring quantifies impairments as percentages, aiding clinical and workplace assessments.
System usability scale (SUS) (applicable for group B) | 3 weeks
  The System Usability Scale (SUS) is a widely used tool for evaluating the perceived usability of products and systems. It consists of a 10-item questionnaire using a 5-point Likert scale. The SUS provides a quick, reliable method to assess user satisfaction and ease of use for various digital interfaces, including websites, software applications, and hardware devices. It generates a score ranging from 0 to 100, with higher scores indicating better usability.

CONTACTS AND LOCATIONS:
Locations (1):
- Thumbay Medicity, Al Jurf, Ajman, Ajman, United Arab Emirates

IPD SHARING:
Plan to Share IPD: Undecided